CLINICAL TRIAL: NCT02906124
Title: A Multinational Observational Study to Evaluate the Safety of Repatha® in Pregnancy
Brief Title: Study to Evaluate the Safety of Repatha® in Pregnancy
Status: Terminated | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20150162
Record Dates: First submitted 2016-08-01; First posted 2016-09-19 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Hypercholesterolaemia; Pregnancy
Keywords: hypercholesterolaemia; Lipid lowering therapies; Pregnancy
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Repatha® exposed: Females with familial hypercholesterolaemia (FH) exposed to Repatha® in the 15 weeks prior to or during pregnancy or during breastfeeding
- Non exposed to Repatha®: Pregnant females with familial hypercholesterolaemia (FH) not exposed to Repatha® and enrolled into this study, overall and stratified by lipid lowering therapy use

SUMMARY:
To evaluate pregnancy and infant outcomes among females diagnosed with familial hypercholesterolaemia (FH), exposed to Repatha® during pregnancy. This includes follow-up of their infants to the age of 12 months

DETAILED DESCRIPTION:
Women diagnosed with familial hypercholesterolaemia (FH), treated at centres in Europe, South Africa and Australia, with pregnancy confirmed during the study observation period and who provide informed consent to participate in the study.

Exposed subjects are women who received Repatha® during pregnancy and/or breastfeeding; unexposed subjects are women who have not received Repatha® during pregnancy and/or breast-feeding. In infants, exposure may occur in utero and/or via breast milk, within 15 weeks following the date of Repatha® dosing in the mother

ELIGIBILITY:
Inclusion Criteria:

* Females diagnosed with Familial hypercholesterolaemia (FH).
* Confirmed pregnancy during the study observation period.
* Pregnancies identified retrospectively but within the study period will be included
* Multiple pregnancies, occurring in the same woman within the study period, will all be included (as separate pregnancies)
* Provided informed consent to follow-up in this study, for subject and their infant(s) born during the study observation period

Exclusion Criteria:

There are no exclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sites in Europe, South Africa and Australia where pregnant familial hypercholesterolaemia (FH) Patients are treated with and without Repatha®
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Any incident of congenital anomaly | From birth up to 12 months of age
  Any incidence of congenital anomaly recorded on the study specific eCRF

SECONDARY OUTCOMES:
End product of pregnancy summarised within 3 main categories: Fetal death, termination of pregnancy and live birth | From pregnancy diagnosis through to birth
  Live birth(s), still birth, spontaneous loss, elective termination, ectopic pregnancy, complication of pregnancy (pre-eclampsia, gestational diabetes)
Status of infant at delivery | At delivery
  Collection of data on gender; gestational age; Apgar score and birth weight
Details of any hospitalisations of infant, documented from delivery to 12 months of age. | From delivery to 12 months of age
  Collection of hospitalisation reason, admission and discharge dates.
Mode of delivery of infant | At delivery
  Collection of delivery mode classified by caesarian section, normal vaginal delivery, operative vaginal delivery and vaginal breech delivery
Growth of infant at 6 months post delivery | Between birth and 6 months of age
  Data on infant growth measured by weight in kilograms.
Details of any chronic medication taken by infant from birth to 12 months of age | From birth to 12 months of age
  Details of any chronic medication prescribed to infant from birth to 12 months of age
Developmental milestones measured at 6 and 12 months of age | At 6 and 12 months of age of infant
  A check of developmental milestones made at 6 and 12 months of age. Details collected where expected milestones were not met.
Details of any complication of delivery | At delivery
  Recording the occurence of any complications of delivery as listed; requirement for blood transfusion, thromboembolism, fetal distress and amniotic fluid abnormality
Growth of infant at 12 months post delivery | Between birth and 12 months of age
  Data on infant growth measured by weight in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (47):
- Australia (2):
  - Research Site, Camperdown, New South Wales
  - Research Site, Clayton, Victoria
- Research Site, Graz, Austria
- Belgium (5):
  - Research Site, Aalst
  - Research Site, Edegem
  - Research Site, La Louvière
  - Research Site, Leuven
  - Research Site, Liège
- Czechia (4):
  - Research Site, Hradec Králové
  - Research Site, Liberec
  - Research Site, Prague
  - Research Site, Uherské Hradiště
- Research Site, Aarhus N, Denmark
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Piraeus
- Italy (12):
  - Research Site, Cagliari
  - Research Site, Cinisello Balsamo (MI)
  - Research Site, Ferrara
  - Research Site, Genova
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Roma
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
- Research Site, Oslo, Norway
- Research Site, Bratislava, Slovakia
- Spain (5):
  - Research Site, Córdoba, Andalusia
  - Research Site, Málaga, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Reus, Catalonia
- Sweden (2):
  - Research Site, Malmo
  - Research Site, Uppsala
- Switzerland (2):
  - Research Site, Geneva
  - Research Site, Reinach
- United Kingdom (5):
  - Research Site, Bournemouth
  - Research Site, Cambridge
  - Research Site, Manchester
  - Research Site, Peterborough
  - Research Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com